CLINICAL TRIAL: NCT01578603
Title: Effects of Two Sugar Substituted Chewing Gums Plus Tooth Brushing on Different Caries and Gingivitis Related Variables: a Double Blind, Randomized Controlled Clinical Trial
Brief Title: Effects of Two Sugar Substituted Chewing Gums on Caries and Gingivitis Variables
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, María Cecilia Martínez-Pabón, Profesora Asociada, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 15-2010
Record Dates: First submitted 2012-04-09; First posted 2012-04-17 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Dental Plaque; Saliva Altered; Gingivitis
Keywords: prevention & control; Xylitol; casein phosphopeptide amorphous calcium phosphate complex; Streptococcus mutans; saliva; dental plaque; gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis | interventions — Xylitol; Sugar Alcohols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sugar substituted chewing gum A (Experimental)
  Interventions: Dietary Supplement: casein phosphopeptide amorphous calcium phosphate complex
- Sugar substituted chewing gum B (Experimental)
  Interventions: Dietary Supplement: xylitol

INTERVENTIONS:
Dietary Supplement: xylitol — 6 g/day, for a month, by chewing 2g three times daily after meals.
  Other Names: sugar alcohol
  Arms: Sugar substituted chewing gum B
Dietary Supplement: casein phosphopeptide amorphous calcium phosphate complex — two pieces of the commercial presentation three times daily after meals
  Other Names: CPP-ACP complex
  Arms: sugar substituted chewing gum A

SUMMARY:
The purpose of this study is to determine the effect of three times a day mastication, during a follow-up period of 4 weeks, of two sugar-substituted chewing gums on various factors associated with dental caries and gingivitis.

DETAILED DESCRIPTION:
The purpose of this paper is to compare the effect of daily consumption of two sugar-free chewing gum, one with Recaldent and one with Xylitol, added to traditional hygiene (brushing, fluoridated toothpaste and dental floss), in clinical features such as the accumulation of plaque and gingival inflammation, microbiological characteristics of saliva as the counts of cariogenic microorganisms and facultative anaerobes, and some physicochemical properties of saliva such as pH and concentrations of calcium and inorganic phosphate.

To this there was a general call among dental students at the University of Antioquia and those who expressed their intention to participate voluntarily with informed consent, were examined clinically and randomly assigned to one of the study groups (Recaldent or Xylitol) or the control group.

After a month of baseline examination and the daily use of the same instruments of oral hygiene and chewing of 6 pellets of each chewing gum (in the case of study groups), all variables are re-examined.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* dental student

Exclusion Criteria:

* less than 26 teeth in mouth
* use of orthodontic appliances
* use of antibiotics the last 3 months

Ages: 16 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Turesky index | a month
  dental plaque assessment

SECONDARY OUTCOMES:
Gingival index | a month
  gingival inflammation
salivary pH | a month
Streptococcus mutans | a month
  number of Streptococcus mutans in saliva
Ca levels | a month
  levels of calcium in saliva
facultative microorganisms | a month
  number of facultative microorganisms in saliva
Lactobacillus | a month
  levels of Lactobacillus spp. in saliva
phosphate levels | a month
  inorganic phosphate leves in saliva
BOP index | a month
  bleeding on probing

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Martínez-Pabón, MsC Microb, Study Director — Universidad de Antioquia
Locations (1):
- Facultad de Odontología, Universidad de Antioquia, Medellín, Antioquia, Colombia